CLINICAL TRIAL: NCT01982214
Title: Effects of Whole Body Vibration (WBV) on Musculoskeletal System of Aged Women
Acronym: VIBROS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Association pour le Développement de la Recherche sur l'Appareil Locomoteur dans la Loire (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0908095; 2009-A00896-51 (Other: ANSM)
Record Dates: First submitted 2013-11-06; First posted 2013-11-13 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-08

CONDITIONS: Osteopenia
Keywords: osteopenia; whole body vibration; women; bone microarchitecture; bone density
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- sedentary (Sham Comparator): No intervention
  Interventions: Device: sedentary
- Vibration (Experimental): Subjects in this group will be submitted to the WBV for 5 to 20 minutes, 2 or 3 times a week while 12 months. The training included light squats at 35-50 Hz and ended up by stretching and relaxation exercises.
  Interventions: Device: Vibration

INTERVENTIONS:
Device: sedentary — No intervention
  Arms: sedentary
Device: Vibration — Subjects will be submitted to the WBV for 5 to 20 minutes, 2 or 3 times a week with frequencies between 35 to 50 Hz while 12 months
  Other Names: Power Plate Limited, London, UK
  Arms: Vibration

SUMMARY:
A controlled, non-randomized trial will be carried out in 240 postmenopausal women, aged 55-75 years, over a 18-month period. The group 1 received a physical intervention, consisting of whole body vibration (WBV) over 12 months followed by training arrest during 6 months. The group 2 served as sedentary control. WBV training is performed 2 or 3 times per week, with each session lasting 20 minutes. The training included light squats at 35-50 Hz and ended up by stretching and relaxation exercises at 50 Hz. Bone, muscle and postural evaluations will be performed at the beginning, 6, 12 and 18 months in each group with evaluation of bone micro-architectural trabecular and cortical compartments, at the weight bearing tibia and the non weight bearing radius.

The primary outcome of the project is the pre, mid, and post evaluations of bone. Bone exploration included dual x-ray absorptiometry (DXA) and high resolution peripheral quantitative computed tomography (HR-pQCT). Bone Mass Density (BMD) will be evaluated by DXA at lumbar, femoral levels and humeral, macro and micro-architectures of the cortical and trabecular compartments will be evaluated in distal radius and tibia by HR-pQCT and bone markers will be analyzed longitudinally. The secondary aim is to assess muscle performance and proprioception. Finally will be assessed markers of cartilage degradation and synthesis, no study has been published on this tissue.

ELIGIBILITY:
Inclusion Criteria:

* Be sedentary (less than 2 hours physical activity of low intensity per week)
* Fracture risk Densitometry Risk factors (FRAX) index between 3 and 10%
* Consent form signed

Exclusion Criteria:

* Bone concomitant disease (such as Paget's disease, osteomalacia),
* Endocrinopathy defined on biological criteria (such as Cushing's disease, hyperparathyroidism, hyperthyroidism, hypogonadism),
* Smoking habits (more than 5 cigarettes per day), chronic alcoholism,
* Treatments received in the previous 6 months affecting bone metabolism such as anabolics, anti-osteoporotic treatment, corticosteroids.
* Having a prosthesis (femur and knee),or recently placed metal bouts or plates
* acute thrombotic problems,
* severe heart- and vascular diseases,
* recent injuries due to operation or polyclinical intervention,
* acute hernia, discopathy, spondylolysis,
* epilepsy,
* severe migraine,
* pacemaker,
* every neurodegenerative or neuromuscular disease,
* dementia

Ages: 55 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2010-04; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Trabecular bone volume at the femoral neck | 12 month
  bone densitometric parameters will be evaluated with DXA (dual x-ray absorptiometry)

SECONDARY OUTCOMES:
Serum bone markers | 12 month
  We will evaluated the activity of bone serum markers of bone formation (amino-terminal propeptide type I procollagen, PINP) and of bone resorption (C telopeptide of type I collagen, S-CTX).
Bone cortical compartment at radius and tibia | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Thierry THOMAS, MD PhD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France